CLINICAL TRIAL: NCT00445315
Title: A Phase 1, Randomized, Double Blind (3rd Party Open), Placebo-controlled, Sequential Group, Multicentre Study To Evaluate The Multiple Dose Safety, Tolerability, Pharmacokinetics And Pharmacodynamics, of PF-00868554 in Hepatitis C Virus (HCV) Positive Otherwise Healthy Patient Volunteers
Brief Title: A Phase 1 Study Of PF-00868554 In Hepatitis C Virus (HCV) Positive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: A8121002
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — filibuvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 2 (Experimental)
  Interventions: Drug: PF-00868554
- 3 (Experimental)
  Interventions: Drug: PF-00868554
- 1 (Experimental)
  Interventions: Drug: PF-00868554
- 4 (Experimental)
  Interventions: Drug: PF-00868554
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-00868554 — 300 mg BID
  Arms: 1
Drug: PF-00868554 — 450 mg BID
  Arms: 2
Drug: PF-00868554 — 100 mg BID
  Arms: 3
Drug: PF-00868554 — 300 mg TID
  Arms: 4
Drug: Placebo — Placebo
  Arms: 5

SUMMARY:
Assess the safety, tolerability and pharmacokinetics of multiple oral doses of PF-00868554 in HCV positive patient volunteers

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA ≥ 100,000 IU/mL at screening
* Genotype 1a or 1b

Exclusion Criteria:

* Current or prior treatment with IFN and/or RBV
* Evidence of decompensated liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Brussels, Belgium
- Pfizer Investigational Site, Berlin, Germany
- Pfizer Investigational Site, Dundee, United Kingdom

REFERENCES:
- [Derived] Wagner F, Thompson R, Kantaridis C, Simpson P, Troke PJ, Jagannatha S, Neelakantan S, Purohit VS, Hammond JL. Antiviral activity of the hepatitis C virus polymerase inhibitor filibuvir in genotype 1-infected patients. Hepatology. 2011 Jul;54(1):50-9. doi: 10.1002/hep.24342. PMID 21488067
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8121002&StudyName=A%20Phase%201%20Study%20Of%20PF-00868554%20In%20Hepatitis%20C%20Virus%20%28HCV%29%20Positive%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-00868554 100 mg Twice Daily: PF-00868554 100 milligram (mg) powder for oral solution, twice daily on Day 1 through Day 7 and once in morning on Day 8.
- PF-00868554 300 mg Twice Daily: PF-00868554 300 mg powder for oral solution, twice daily on Day 1 through Day 7 and once in morning on Day 8.
- PF-00868554 300 mg Three Times Daily: PF-00868554 300 mg powder for oral solution, three times daily on Day 1 through Day 7 and once in morning on Day 8.
- PF-00868554 450 mg Twice Daily: PF-00868554 450 mg powder for oral solution, twice daily on Day 1 through Day 7 and once in morning on Day 8.
- Placebo: Placebo matched to PF-00868554 powder for oral solution, twice daily or three times daily on Day 1 through Day 7 and once in morning on Day 8.
Period: Overall Study
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily | Placebo
Started | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Customized [Number; unit: participants]
  18 to 44 years | 3 | 2 | 2 | 4 | 6 | 17
  45 to 64 years | 3 | 4 | 3 | 2 | 2 | 14
  greater than or equal to 65 years | 0 | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 1 | 1 | 5
  Male | 6 | 5 | 4 | 5 | 7 | 27

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax): Day 1
Time Frame: 0 hours (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 hours post-dose for twice daily dose; 0 hours (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 hours post-dose for three times daily dose
Population: Per Protocol (PP) analysis set included all participants who received PF-00868554 and had sufficient plasma concentration data to enable calculation of the pharmacokinetics (PK) parameters.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 3467.0 (1085.36) | 27437.1 (7875.45) | 23046.7 (10526.66) | 48392.6 (13466.65)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax): Day 8
Time Frame: 0 hours (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 hours post-dose
Population: PP analysis set included all participants who received PF-00868554 and had sufficient plasma concentration data to enable calculation of the PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 5858.8 (2312.65) | 33111.4 (8680.94) | 30919.1 (6576.52) | 57724.5 (17739.87)

3. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax): Day 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour | 1.00 [0.50 to 1.50] | 0.50 [0.50 to 1.00] | 0.51 [0.50 to 1.00] | 0.50 [0.50 to 1.03]

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax): Day 8
Time Frame: 0 hours (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour | 0.76 [0.50 to 1.00] | 0.50 [0.50 to 1.00] | 0.50 [0.48 to 0.50] | 0.50 [0.48 to 0.52]

5. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau): Day 1
Description: Area under the plasma concentration time-curve from time zero to end of dosing interval (tau), where dosing interval is 8 hours for three times daily regimens and 12 hours for the twice daily regimens.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hour/mL | 13816.6 (6698.11) | 73653.0 (19681.78) | 52933.7 (30925.32) | 110158.1 (44416.51)

6. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau): Day 8
Description: as for outcome 5
Time Frame: 0 hours (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hour/mL | 20632.5 (13934.95) | 84983.3 (20225.45) | 59492.4 (26992.82) | 120849.4 (42396.74)

7. Primary Outcome: Minimum Observed Plasma Trough Concentration (Cmin): Day 8
Description: The Cmin of PF-04691502 was assessed following repeated oral dose administration for 8 days (multiple dose PK).
Time Frame: 0 hours (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 hours post-dose on Day 8
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 448.6 (422.18) | 904.8 (342.73) | 1055.9 (437.59) | 706.0 (661.12)

8. Primary Outcome: Plasma Decay Half-Life (t1/2): Day 8
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. The t1/2 of PF-04691502 was assessed following repeated oral dose administration for 8 days (multiple dose PK).
Time Frame: 0 hours (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 hours post-dose on Day 8
Population: PP analysis set included all participants who received PF-00868554 and had sufficient plasma concentration data to enable calculation of the PK parameters. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 5 | 6 | 6
hour | 12.58 (3.01) | 10.77 (4.29) | 9.17 (0.62) | 8.13 (0.72)

9. Primary Outcome: Observed Accumulation Ratio (Rac)
Description: Rac was calculated as, area under the curve from time zero to end of dosing interval on Day 8 (AUCtau) divided by area under the curve from time zero to end of dosing interval on Day 1(AUCtau).
Time Frame: 0 hours (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 hours post-dose on Day 1; 0 hours (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 hours post-dose on Day 8
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6 | 6
ratio | 1.49 (0.25) | 1.15 (0.24) | 1.12 (0.15) | 1.09 (0.19)

10. Primary Outcome: Observed Accumulation Ratio for Cmax (Rac Cmax)
Description: Rac Cmax was calculated as, maximum observed plasma concentration on Day 8 (Cmax) divided by maximum observed plasma concentration on Day 1(Cmax).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6 | 6
ratio | 1.68 (0.46) | 1.20 (0.25) | 1.34 (0.28) | 1.19 (0.46)

11. Primary Outcome: Cumulative Amount of Drug Recovered Unchanged in Urine (Ae): Day 1
Description: Ae is the cumulative amount of drug recovered unchanged in urine during the dosing interval, where the dosing interval is 12 hours. Cumulative amount was calculated as sum of urine drug concentration in sample volume for each collection interval. Sample volume = (urine weight in gram [g]/1.020), where 1.020 g/mL is the approximate specific gravity of urine.
Time Frame: 0 to 12 hours, 12 to 24 hours post-dose
Population: PP analysis set included all participants who received PF-00868554 and had sufficient plasma concentration data to enable calculation of the PK parameters. Urine collection interval was 12 hours and not 8 hours; therefore, urinary PK parameters were not calculated for three times daily regimens.
Measure: Geometric Mean (Standard Deviation); unit: nanogram
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6
nanogram | 13490943.6 (5465341.72) | 47306427.2 (10029440.68) | 58500433.1 (23166241.78)

12. Primary Outcome: Cumulative Amount of Drug Recovered Unchanged in Urine (Ae): Day 8
Description: as for outcome 11
Time Frame: 0 to 12 hours, 12 to 24 hours post-dose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: nanogram
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6
nanogram | 23157156.8 (8370778.62) | 61249508.4 (13917200.98) | 59663120.9 (17455075.93)

13. Primary Outcome: Percent of Dose Recovered Unchanged in Urine (Ae%): Day 1
Description: Percent of dose recovered unchanged in urine during the dosing interval=100*(cumulative amount of drug recovered unchanged in urine [Ae] divided by dose), where the dosing interval is 12 hours.
Time Frame: 0 to 12 hours, 12 to 24 hours post-dose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: percent dose recovered
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6
percent dose recovered | 13.49 (5.46) | 15.77 (3.34) | 13.00 (5.15)

14. Primary Outcome: Percent of Dose Recovered Unchanged in Urine (Ae%): Day 8
Description: Percent of dose recovered unchanged in urine during the dosing interval=100 (cumulative amount of drug recovered unchanged in urine [Ae] divided by dose), where the dosing interval is 12 hours.
Time Frame: 0 to 12 hours, 12 to 24 hours post-dose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: percent dose recovered
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6
percent dose recovered | 23.16 (8.37) | 20.42 (4.64) | 13.26 (3.88)

15. Primary Outcome: Renal Clearance (CLr): Day 1
Description: Renal clearance was calculated as cumulative amount of drug recovered unchanged in urine during the dosing interval (Ae) divided by area under the plasma concentration time-curve from time zero to end of dosing interval (AUCtau), where dosing interval is 12 hours.
Time Frame: 0 to 12 hours, 12 to 24 hours post-dose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: mL/minute
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6
mL/minute | 16.27 (6.50) | 10.70 (2.19) | 8.85 (5.90)

16. Primary Outcome: Renal Clearance (CLr): Day 8
Description: as for outcome 15
Time Frame: 0 to 12 hours, 12 to 24 hours post-dose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: mL/minute
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 450 mg Twice Daily
Number analyzed (Participants) | 6 | 6 | 6
mL/minute | 18.70 (3.79) | 12.01 (3.50) | 8.23 (4.26)

17. Primary Outcome: Ratio of 6 Beta-Hydroxyl Cortisol to Cortisol: Day 1
Description: Urine 6 beta-hydroxyl cortisol and cortisol concentrations were measured using high performance liquid chromatography-tandem mass spectrometry (HPLC-MS/MS).
Time Frame: -24 to 0 hours (pre-dose) on Day 1 (Day 0)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
ratio | 2.93 (1.55) | 3.94 (1.42) | 4.65 (2.95) | 4.32 (1.62) | 3.56 (1.68)

18. Primary Outcome: Ratio of 6 Beta-Hydroxyl Cortisol to Cortisol: Day 8
Description: as for outcome 17
Time Frame: 0 to 24 hours post-dose on Day 8
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
ratio | 3.79 (1.47) | 3.90 (1.56) | 5.26 (2.79) | 4.58 (0.97) | 4.30 (1.05)

19. Primary Outcome: Day 8 to Day 1 Ratio of the 6 Beta-Hydroxyl Cortisol to Cortisol Ratios
Description: as for outcome 17
Time Frame: -24 to 0 hours (pre-dose) on Day 1 (Day 0); 0 to 24 hours post-dose on Day 8
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
ratio | 1.29 (0.38) | 0.99 (0.24) | 1.13 (0.09) | 1.06 (0.27) | 1.20 (0.62)

20. Secondary Outcome: Change From Baseline in Plasma Log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Viral Load at Day 8
Description: HCV RNA levels were determined using the Abbott RealTime HCV polymerase chain reaction (PCR) assay (lower limit of detection [LOD] = 12 international unit per milliliter [IU/mL]). Baseline value calculated as the average of the screening Day 0 and Day 1 pre-dose measurements. The plasma HCV RNA data was log10 transformed, and the change in log10 HCV RNA at Day 8 post-dose from baseline was calculated.
Time Frame: Baseline, Day 8
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
log10 copies/mL
  Baseline | 6.14 (0.39) | 6.05 (0.35) | 6.02 (0.50) | 5.75 (0.65) | 6.02 (0.58)
  Change at Day 8 | -0.68 (0.38) | -1.26 (0.58) | -1.95 (0.51) | -1.21 (0.70) | -0.08 (0.10)

21. Secondary Outcome: Number of Participants With Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Variants Resistant to PF-00868554
Time Frame: Screening up to Day 8
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
participants | 0 | 6 | 2 | 3 | 0

ADVERSE EVENTS:
Arm/Group | PF-00868554 100 mg Twice Daily | PF-00868554 300 mg Twice Daily | PF-00868554 300 mg Three Times Daily | PF-00868554 450 mg Twice Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 5/6 | 5/6 | 3/6 | 5/6 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00868554 100 mg Twice Daily (N=6) | PF-00868554 300 mg Twice Daily (N=6) | PF-00868554 300 mg Three Times Daily (N=6) | PF-00868554 450 mg Twice Daily (N=6) | Placebo (N=8)
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1
Foreign body sensation in eyes (Eye disorders) | 1 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Application site erythema (General disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 2
Liver tenderness (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 2 | 3
Intercostal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Designation of outcomes as primary, secondary based on team's input. Results for relationship analyses of baseline susceptibility to PF-00868554 and/or non-structural 5B genotype and change in HCV RNA was not done, as per change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.